CLINICAL TRIAL: NCT06808711
Title: Evaluation of the Tolerance and Effectiveness of Buccocean Mouthwash Under Real-use Conditions
Brief Title: Usage Test on a New Cosmetic Product: Mouthwash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YSLab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BUCCOCEAN
Record Dates: First submitted 2025-01-23; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Sensitive Gum; Gum Inflammation
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buccocéan (Experimental): Mouthwash, twice a day
  Interventions: Other: Buccocéan mouthwash
- Marketed mouthwash (Active Comparator): Mouthwash, twice a day
  Interventions: Other: Marketed mouthwash

INTERVENTIONS:
Other: Buccocéan mouthwash — Normal conditions of use
  Arms: Buccocéan
Other: Marketed mouthwash — Normal conditions of use
  Arms: Marketed mouthwash

SUMMARY:
The goal of this clinical trial is to learn if a new mouthwash can help soothing oral mucosa in adult patients with sensitive gums. The main questions it aims to answer are:

* Does the investigated mouthwash soothe red gum?
* Has the mouthwash antibacterial activities? Researchers will compare with a marketed mouthwash to see if the observed effect is due to the formula or to the general rinsing effect of any mouthwash.

Participants will be asked to use the investigated mouthwash or the comparative mouthwash twice a day for 21 days.

DETAILED DESCRIPTION:
Severity of gingival inflammation is evaluated using the Loë & Silness scale, which includes 4 scores (0=no inflammation, 3=Significant inflammation, redness, accentuated hypertrophy with spontaneous hemorrhagic tendency and ulceration) by the dentist, on Day 0 and on Day 7.

Presence of dental plaque is evaluated using the Loë & Silness scale, which includes 4 scores (0=no dental plaque, 3=Abundant plaque along the gingival margin; the spaces between the teeth are filled with plaque) by the dentist, on Day 0 and on Day 7.

Changes in the gingival microbiota is evaluated through the analysis of bacteria on D0 and D7 by swab sampling on the occlusal and buccal surfaces at the gum line.

Tolerance (adverse effects) will also be studied by recording any adverse effect.

ELIGIBILITY:
Inclusion Criteria:

* Person (man, woman) aged 18 or over,
* Person with a gingival index ≥ 2 (according to Loë & Silness) on at least 10% of teeth (i.e. 3 teeth) at the inclusion visit
* Person capable of following the instructions for using the product,
* Person agreeing to come for a dental consultation 7 days (+/- 1 day) after the inclusion visit,
* Volunteer informed and having signed their informed consent form,
* Volunteer person affiliated to a social security scheme (Art L1121-11 of the CSP).

Exclusion Criteria:

* Person who has regularly used mouthwash in the last month,
* Person suffering from periodontitis
* Person having a scaling treatment planned in the session, or having had a scaling treatment in the 6 months preceding the inclusion visit,
* Person having had antibiotic or antifungal treatment in the 3 months preceding the visit,
* Person taking anti-coagulant or anti-aggregant or immunosuppressive or anti-cancer treatment (chemotherapy or radiotherapy of the head and neck)
* Person at risk of infective endocarditis,
* Person with a known sensitivity or allergy to one of the components of mouthwashes, including components derived from essential oils (Eucalyptol, thymol, menthol, limonene).
* Volunteer participating in intervention research.
* Vulnerable people referred to in articles L. 1121-5 to 8 and L. 1122-1-2 of the Public Health Code (institutionalized volunteers, deprived of their liberty or placed under legal protection (guardianship or curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Tolerance of the product | From enrollment to the end of treatment at 3 weeks
  Tolerance of the mouthwash expressed by the number of adverse effects linked to the product

SECONDARY OUTCOMES:
Soothing effect on irritated gums | At Day 0 and Day 7
  Gingival index assessed by the dentist (Grade 0-3)
Effect on dental plaque | At Day 0 and Day 7
  Plaque index by the dentist (grade 0-3)
Effect on the oral microbiota | At Day 0 and Day 7
  Evaluation of the gingival microbiota by swab sampling on the occlusal and buccal surfaces at the gum line

CONTACTS AND LOCATIONS:
Locations (1):
- Dentistry center, Rennes, France